CLINICAL TRIAL: NCT05085054
Title: Induction Therapy With Targeted Therapy Followed by Surgery for Stage IIIB and IV Non-small Cell Lung Cancer: a Multi-center, Single-arm, Prospective Clinical Study
Brief Title: Salvage Surgery Following Downstaging of Advanced Non-small Cell Lung Cancer by Targeted Therapy (SDANT)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDANT
Record Dates: First submitted 2021-09-21; First posted 2021-10-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Unresectable; Advanced NSCLC; Targeted Therapy; Salvage Surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- targeted therapy+salvage surgery (Experimental): Participants treated with targeted therapy without progression and radiological confirmation of tumor downstaging (≤stage IIIA) by PET-CT followed by salvage surgery were enrolled into the group of targeted therapy plus salvage surgery.
  The molecular targeted agents used in our study included osimertinib (80 mg, once a day) . Salvage surgery was defined as surgical intervention based on standard operation (lobectomy plus lymphadenectomy) of NSCLC for advanced patients who initially had no surgical indications, but achieved significant downstaging (≤stage IIIA) without progression after targeted therapy.
  Targeted therapy was continued after salvage surgery until progression.
  Interventions: Drug: Osimertinib Mesylate

INTERVENTIONS:
Drug: Osimertinib Mesylate — Participants will receive targeted therapy followed by salvage surgery

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of neoadjuvant targeted therapy followed by surgery in participants with advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
Advanced non-small cell lung cancer (NSCLC) accounts for a high proportion of lung cancer cases. Targeted therapy improve the survival in these patients, but acquired drug resistance will inevitably occur. If tumor downstaging is achieved after targeted therapy, could surgical resection before drug resistance improve clinical benefits for patients with advanced NSCLC? Here, the investigators conducted a clinical trial showing that for patients with advanced driver gene mutant NSCLC who did not progress after targeted therapy, salvage surgery (SS) could improve progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of NSCLC with confirmed activation of driver gene mutation (EGFR mutant: exon 19 deletion or exon 21 L858R mutation; ALK-rearrangement) by amplification refractory mutation system (ARMS);
* stage IIIB-IV according to the eighth edition of the American Joint Committee on Cancer staging system confirmed by pathological diagnosis and positron emission tomography-computed tomography (PET-CT) and biopsy
* Written informed consent provided；
* Age 18-70 when signing the consent form, both male and female;
* The ECOG score is 0 or 1;
* Adequate hematological function, liver function and renal function;
* Female participants should not be pregnant or breast-feeding.

Exclusion Criteria:

* Previously received systemic anti-tumor therapy for non-small cell lung cancer;
* Subjects who have received chest radiotherapy in the past;
* Known human immunodeficiency virus (HIV) infection;
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease);
* Pregnancy or breast-feeding women;
* Ingredients mixed with small cell lung cancer patients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 3 year
  Progression-Free Survival

SECONDARY OUTCOMES:
OS | 3 year
  Overall Survival
Resectability rate | 1 year
  Resectability rate is defined as the percentage of patients who were able to undergo surgery after neoadjuvant therapy.

IPD SHARING:
Plan to Share IPD: No